CLINICAL TRIAL: NCT05314868
Title: Postmarket, Retrospective Evaluation of Photo-oxidized Decellularized Bovine Pericardium Used as a Patch in Cardiac Repair or Reconstruction Surgery
Brief Title: Retrospective Evaluation of Photo-oxidized Decellularized Bovine Pericardium in Cardiac Repair or Reconstruction Surgery
Acronym: Retro-C
Status: Terminated | Type: Observational
Why Stopped: Sponsor declined to continue funding the study.
Sponsor: Artivion Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHF1901.000-M (11/19)
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease; Cardiac Anomaly
Keywords: bovine pericardium patch; cardiac repair; cardiac reconstruction
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Primary cohort: Pediatrics or adults who underwent cardiac repair surgery that nessecitated the use of a PhotoFix patch.
  Interventions: Device: PhotoFix

INTERVENTIONS:
Device: PhotoFix — Surgical repair with patch.
  Other Names: PhotoFix Decellularized Bovine Pericardium

SUMMARY:
The objective of this postmarket, retrospective, single center study is to evaluate the clinical outcomes of patients who have received PhotoFix® Decellularized Bovine Pericardium (PhotoFix) as a patch within a cardiac surgical repair or reconstruction procedure. PhotoFix is prepared from bovine pericardium, which is stabilized using a dye-mediated photo-oxidation process and sterilized using aseptic processing techniques.

DETAILED DESCRIPTION:
This study will include a review of approximately 300 charts spanning the implant period of January 1, 2018 through June 30, 2019. Those that meet the inclusion and exclusion criteria will undergo full review and data extraction to be captured in the electronic database. Given the retrospective nature of the study design, a Waiver of Consent will be requested from the Institutional Review Board (IRB). Potential subjects this study are pediatrics or adults who underwent cardiac repair surgery that necessitated the use of a patch. Targeted cardiac procedures include intracardiac repair (including annulus and septal repair), great vessel repair (including superior vena cava, inferior vena cava, pulmonary arteries, pulmonary veins, and ascending aorta), and suture line buttressing and pericardial closure. Follow-up data will be abstracted from the subject's medical record. Study specific testing, including imaging and laboratory testing, will not be required.

ELIGIBILITY:
Inclusion Criteria:

* Subject has undergone a cardiac procedure which falls within the indications for use and required the use of PhotoFix Decellularized Bovine Pericardium

Exclusion Criteria:

* Subject required valve leaflet repair using PhotoFix

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Candidates for this study are pediatrics or adults who underwent cardiac repair surgery that necessitated the use of a patch.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
  Mortality

SECONDARY OUTCOMES:
All-cause reoperation | Up to 5 years
  The total number of unplanned reoperations required in patients over the follow-up period, which include the repair or alteration of the surgical area around the patch. Patients with planned reoperations, such as CHD staged surgeries, will not be considered.
Device-related reoperation | Up to 5 years
  The total number of unplanned reoperations required in patients over the follow-up period, which are determined by the surgeon to be device-related.
Explant | Up to 5 years
  The total number of device explants over the course of follow-up.
Morbidity | Up to 5 years
  The total number of any adverse event, with specific focus on cardiovascular complications which have the potential to be device-related.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Baird, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital of Boston, Boston, Massachusetts, United States